CLINICAL TRIAL: NCT05264012
Title: Incidence, Risk Factors and Impact of Significant Pain in Patients Undergoing Neurosurgery
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Sriganesh Kamath, Principal Investigator, National Institute of Mental Health and Neuro Sciences, India
Other Study IDs: 111
Record Dates: First submitted 2022-01-28; First posted 2022-03-03 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain; Neurosurgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Neurosurgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cranial neurosurgery: Patients undergoing cranial neurosurgery
  Interventions: Procedure: Neurosurgery
- Non-cranial neurosurgery: Patients undergoing non-cranial neurosurgery including spine surgery
  Interventions: Procedure: Neurosurgery

INTERVENTIONS:
Procedure: Neurosurgery — Neurosurgery

SUMMARY:
The proposed study intends to evaluate incidence of postoperative pain after neurosurgery. This study is likely to help in understanding of the magnitude of this problem in our country and inform about possible predictors which will help institute pre-emptive interventions to mitigate modifiable risk factors of pain after neurosurgery.

DETAILED DESCRIPTION:
Data regarding potential risk factors for postoperative pain will be collected. Preoperative factors (preoperative pain, anxiety or depression, perception about surgery, age, gender, socio-economic status, educational level, domicile location, obesity, surgical site [infratentorial or supratentorial or cervical, thoracic or lumbar], use of steroids and analgesics), and intraoperative factors (scalp/ESP/caudal block, incision site infiltration, dose of analgesics such as opioids, paracetamol and non-steroidal anti-inflammatory drugs (NSAIDs), co-analgesics such as nitrous oxide, gabapentionoids, dexmedetomidine, magnesium or lignocaine infusion, anti-epileptics, steroids, minimum alveolar concentration (MAC) of inhalational anesthetics, and duration of surgery and anesthesia) that are likely to be associated with occurrence of postoperative pain will be explored along with relationship between acute and persistent postoperative pain and between intraoperative nociception and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* all eligible consecutive consenting adult patients aged > 18 years with preoperative Glasgow Coma Scale (GCS) score of 15 undergoing elective craniotomies and spine surgeries

Exclusion Criteria:

* children, patients with GCS < 15, patients not extubated within 2 hours of end of anesthesia and those who not able to respond to our questions on outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: undergoing elective cranial and non-cranial neurosurgeries
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain using Numerical Rating Scale | on days 1-3 after surgery
  Acute postoperative pain

SECONDARY OUTCOMES:
duration of postoperative hospital stay in days | through hospital stay, an average of 10 days
  duration of postoperative hospital stay in days
postoperative sleep quality using Likert 1-5 scale | Day 2 after surgery
  sleep quality assessment
patient satisfaction using Likert scale 1-5 | Day 2 after surgery
  patient satisfaction assessment using Likert scale 1-5
Persistent postoperative pain using Numerical Rating Scale (NRS) | 3 and 6 months after surgery
  Chronic Postoperative Pain measured using NRS (from 0 to 10, with 0 = no pain and 10 = maximal pain

CONTACTS AND LOCATIONS:
Overall Officials: Sriganesh K, DM, Principal Investigator — National Institute of Mental Health and Neuro Sciences, India
Locations (1):
- National Institute of Mental Health and Neurosciences, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided